CLINICAL TRIAL: NCT04330976
Title: Preventing Excessive Gestational Weight Gain Via Short Mobile Messages in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)
Brief Title: Preventing Excessive Gestational Weight Gain Via Short Mobile Messages in WIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5U54MD008149-09 (NIH)
Record Dates: First submitted 2020-02-28; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Gestational Weight Gain
MeSH Terms: conditions — Gestational Weight Gain | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition and physical activity intervention (Experimental)
  Interventions: Behavioral: Nutrition and physical activity intervention
- Control (Other)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Nutrition and physical activity intervention — Messages sent on nutrition and physical activity in pregnancy
  Arms: Nutrition and physical activity intervention
Behavioral: Control — Messages sent on general health during pregnancy
  Arms: Control

SUMMARY:
The objective of this trial was to investigate the effect of educational short message service (SMS), or text messages, on gestational weight gain (GWG) in a low-income population.

ELIGIBILITY:
Inclusion Criteria:

* 15-20 weeks gestational age and 18 years of age or older at time of recruitment
* body mass index (BMI) of 25-45 kg/m2 in the first trimester
* possession of a cellular phone with the ability to receive text messages without a charge

Exclusion Criteria:

* conditions requiring a special diet
* multiparous pregnancies
* unable to consent to participate
* unwilling to be randomized

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Change between pre-pregnancy weight and last weight taken before delivery | From date of randomization until delivery of child (e.g. up to 25 weeks)
  Total weight gained during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States